CLINICAL TRIAL: NCT07064915
Title: Impact of a Medical-Financial Partnership Intervention on Parent Mental Health, Perinatal Outcomes, and Child Developmental Risk: A Community-Partnered, Multi-Site Randomized Controlled Trial
Brief Title: Impact of a Medical-Financial Partnership Intervention on Parent Mental Health, Perinatal Outcomes, and Child Developmental Risk
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Adam Schickedanz, Assistant Professor of Pediatrics, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UCLA_DHS_MFP_Evolution_2025; 1R01HD115000-01A1 (NIH)
Record Dates: First submitted 2025-07-07; First posted 2025-07-15 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Child Development; Mental Health
Keywords: Medical-Financial Partnership
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Care Control (No Intervention): This arm is the comparison group, which will receive standard prenatal and pediatric care with social needs screening and intervention as provided by the health care team as usual care (no medical-financial partnership intervention).
- Medical-Financial Partnership Intervention - Prenatal & Postnatal (Experimental): This arm is the first experimental group and participants included in this arm will receive the Medical-Financial Partnership intervention beginning in prenatal care and continuing into the postnatal period.
  Interventions: Behavioral: Medical-Financial Partnership Support
- Medical-Financial Partnership Intervention - Postnatal (Experimental): This arm is the second experimental group and participants included in this arm will receive the Medical-Financial Partnership intervention beginning in the postnatal period.
  Interventions: Behavioral: Medical-Financial Partnership Support

INTERVENTIONS:
Behavioral: Medical-Financial Partnership Support — The Medical-Financial Partnership (MFP) intervention will include (at minimum):
  1. A relationship with a trained MFP intervention team member
  2. Establishment of financial and social goals in the initial meeting, with connection to public anti-poverty programs, employment opportunities, and other income supports, among others, as tailored to participant goals
  3. Establishment of an action plan to reach short, medium and long-term goals in core MFP domains
  4. Co-designing with the participant to identify and refine goals and action steps longitudinally
  5. A standard toolkit for access to financial services and public benefits
  Arms: Medical-Financial Partnership Intervention - Postnatal; Medical-Financial Partnership Intervention - Prenatal & Postnatal

SUMMARY:
Poverty and financial stress are key social drivers of health and root causes of worse health beginning in pregnancy, continuing into childhood, and extending over the life course, but clinical tools to address the health impacts of poverty and financial stress are needed. This trial is of a multi-site medical-financial partnership intervention to examine its effect on parent, perinatal, and child outcomes, as well as health care utilization, and family financial and social risk. This pragmatic randomized clinical effectiveness trial will examine the impact of a clinic-based medical-financial partnership intervention beginning either 1) in the newborn period (Intervention Arm 1) or 2) during prenatal care (Intervention Arm 2) versus controls on parent, child, and family/household outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Being an expectant parent (mother or father) who is either 1) receiving prenatal care or 2) their partner is receiving prenatal care at one of the study's prenatal care clinical sites during recruitment
* Intending at the time of recruitment to have their child receive primary pediatric care at one of the of the study's pediatric primary care clinical sites after birth
* Speaking English or Spanish as primary language

Exclusion Criteria:

* Cognitive impairment or any other condition that would prevent participation in the intervention
* Foster parents
* Parent age under 18 at enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Parent Health-Related Quality of Life, including Mental Health Subscale | Through 24 Months of Child Age
  Measured via participant-reported electronic or paper survey via the Patient Reported Outcome Measurement Information System Short Form Global Scale 10 Item Scale (the PROMIS-10; raw scale range 10-50 then T-Scored, with lower values indicating worse outcomes), this continuous measure is calculated based on Likert scale responses to 10 participant-reported questions/prompts. A mental health subscale of four items assesses depression and anxiety symptom burden and can be T-scored in preparation for analyses.
Child Developmental Risk (in Any Domain) - Ages & Stages Questionnaire (ASQ, version 3) Domain Scores | Through 24 months
  Collected via participant reported standardized Ages & Stages Questionnaire Version 3 (ASQ-3; each domain scale score ranging from 0-60 with threshold cutoffs for delays varying by child age, with lower values indicating a higher likelihood of developmental delay) forms on electronic surveys (preferred source) and at every well child visit beyond age 6 months. The presence of child developmental risk in any of five developmental domains (communication/speech/language, personal-social skills, gross motor skills, fine motor skills, or problem solving) will be measured at well child visits on parent-completed ASQ forms as well as every 6 months via online surveys from child age 6 to 24 months and rates of positive screens for developmental delay will be compared.
Public Benefits Program Enrollment | Through 24 months of child age
  Rates of any public benefits enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Schickedanz, MD PhD, Principal Investigator — University of California, Los Angeles
Locations (4):
- United States (4):
  - Lomita Family Health Center, Harbor City, California
  - Martin Luther King, Jr. Outpatient Center, Los Angeles, California
  - Olive View-UCLA/ERI, Sylmar, California
  - Harbor-UCLA/Lundquist Institute, Torrance, California

IPD SHARING:
Plan to Share IPD: Yes
We plan to share data as required by sponsor policy.
Supporting Information: Study Protocol
Time Frame: After the end of the study or publications, as required by sponsor.